CLINICAL TRIAL: NCT02812498
Title: Teleconsultation in Type 1 Diabetes Mellitus
Acronym: TELEDIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 535-B-102014
Record Dates: First submitted 2016-06-16; First posted 2016-06-24 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: teleconsultation; insulin therapy; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teleconsultation (Experimental): Teleconsultation for patients affected by type 1 diabetes mellitus
  Interventions: Other: Teleconsultation
- Control (Other): Standard visit in outpatient clinic for the same type of patients
  Interventions: Other: Standard

INTERVENTIONS:
Other: Teleconsultation — The patients in the consultation group arranged their bookings on a website, where they could also access to web educational courses or to nutritional and psychological counselling
  Arms: Teleconsultation
Other: Standard — Group of patients followed in a traditional way
  Arms: Control

SUMMARY:
The purpose of this study is to compare the effects on glycemic control of Teleconsultation versus standard visit in outpatient clinic for patients affected by type 1 diabetes mellitus.

DETAILED DESCRIPTION:
The growing incidence of diabetes and the need to contain health care costs empower the necessity to identify new models to cope with regular periodic follow up of patients affected by diabetes mellitus. Telemedicine offers an acknowledged instrument to provide clinical health care at a distance, increasing patient compliance and the achievement of therapeutical goals. This study wants to verify the feasibility and the efficacy of teleconsultation in patients with type 1 diabetes mellitus. In particular by a randomized controlled approach the effects on glycemic control of patients followed by teleconsultation or traditionally in standard visit in the outpatient clinic. The patients in the teleconsultation group will arrange their bookings on a website (http://www.telediabete-fid.it/) In this website they could also access to web educational courses (mainly nutrition, insulin management, glucose monitoring auto-control) or to nutritional and psychological counselling.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by type 1 diabetes mellitus, 5-50 years old under multi injection insulin therapy or under continuous subcutaneous insulin infusion
* with a feasible web access

Exclusion Criteria:

* without a feasible web access
* that need a periodic physical examination

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin HbA1c | 12th month
  HbA1c is the main parameter representing the overall glycemic control. HbA1c can be assessed on three month bases but the value at 12 month is more representative of a sustained effect of this new approach

SECONDARY OUTCOMES:
HbA1c glycosylated hemoglobin | 3rd to 6th to 9th month
  changes of HbA1c glycosylated hemoglobin values
Patient satisfactory assessment by a questionnaire on their perception of advantages (diabetes management, comfort and convenience) and limits (technical problems, poor interaction with physicians) of the service | 12th month
  A score of 1 (low) to 5 (High) will be used
Cost analysis by patient estimation through a questionnaire of the overall cost and time saved thanks to the service | 12th month
  The average amount of cost and time saved will be calculated

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - AO Ospedale Civile Legnano Legnano, Legnano
  - ASST Grande Ospedale Metropolitano Niguarda, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bertuzzi F, Stefani I, Rivolta B, Pintaudi B, Meneghini E, Luzi L, Mazzone A. Teleconsultation in type 1 diabetes mellitus (TELEDIABE). Acta Diabetol. 2018 Feb;55(2):185-192. doi: 10.1007/s00592-017-1084-9. Epub 2017 Dec 5. PMID 29209814